CLINICAL TRIAL: NCT00841958
Title: Efficacy of the Endocardial Stem Cells Implantation in Ischemic Heart Failure Patients
Brief Title: Endocardial Stem Cells Approach Efficacy
Acronym: ESCAPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCVM-029; RU002 (Other: State Research Institute of Circulation Pathology)
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Autologous bone marrow mononuclear stem cells or peripheral blood stem cells — Cells concentration is 150х106 cells/ml (2ml) with CD34+ cells=2.5±1.44%

SUMMARY:
The primary objective of this study is to test that endocardial stem cells implantation in patients who have CAD, low ejection fraction and signs of HF without possibility of CABG and PCI or despite on previous revascularization improves long-term survival compared to MED alone

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are not of childbearing potential
* Age 21-75 years.
* Patients with CAD, NYHA and CCS angina III-IV functional class
* LVEF less than 35% measured by echocardiography or SPECT within three months of study entry
* Unsuitable for initial or repeated conventional revascularization (CABG or PCI)

Exclusion Criteria:

* Failure to provide informed consent.
* Plan for PCI or CABG.
* Non-cardiac illness with a life expectancy of less than 3 year.
* Conditions/circumstances likely to lead to poor treatment adherence (e.g., history of poor compliance, alcohol or drug dependency, psychiatric illness, no fixed abode).
* Previous heart, kidney, liver, or lung transplantation.
* Current participation in another clinical trial in which a patient is taking an investigational drug or receiving an investigational medical device.
* Recent acute myocardial infarction (AMI) within 90 days of study entry
* Successful coronary revascularization (СABG or PCI) within 12 months of study enrollment
* History of moderate to severe aortic stenosis or prosthetic aortic valve
* Permanent atrial fibrillation
* Thrombosis in LV, based on echocardiography data

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2007-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Null Hypothesis (Ho): There is no survival benefit in the stem cells group compared to the control group ( isolate MED therapy). H0: Ө ≤ 1 Alternative Hypothesis (Ha): There is a survival benefit in the stem cells group. HA: Ө > 1 | 2007-2010

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny A Pokushalov, MD, PhD, Principal Investigator — State Research Institute of Circulation Pathology
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- [Result] Pokushalov E, Romanov A, Chernyavsky A, Larionov P, Terekhov I, Artyomenko S, Poveshenko O, Kliver E, Shirokova N, Karaskov A, Dib N. Efficiency of intramyocardial injections of autologous bone marrow mononuclear cells in patients with ischemic heart failure: a randomized study. J Cardiovasc Transl Res. 2010 Apr;3(2):160-8. doi: 10.1007/s12265-009-9123-8. Epub 2009 Sep 24. PMID 20560030
- See also: State Research Institute of Circulation Pathology Official Site — http://www.meshalkin.ru/